CLINICAL TRIAL: NCT02647398
Title: Randomized Study Comparing Two Strategies of Physical Activity in Long-term Breast and Colon Cancer Survivors and Their Impact on Fatigue
Brief Title: Study Comparing Two Strategies of Exercise in Breast and Colon Cancer Survivors and Their Impact on Fatigue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Puerta de Hierro University Hospital (Other)
Collaborators: Universidad Europea de Madrid (Other)
Responsible Party: Principal Investigator, Ana Ruiz-Casado, MD PhD, Puerta de Hierro University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PH-UEM-04
Record Dates: First submitted 2016-01-03; First posted 2016-01-06 (Estimated); Last update posted 2018-04-06 (Actual); Status verified 2018-04

CONDITIONS: Neoplasms; Fatigue
Keywords: Cancer survivors; training; exercise; cancer-related fatigue
MeSH Terms: conditions — Neoplasms; Fatigue; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A: Supervised combined training (Experimental): INTERVENTION: Two supervised 75 min-vigorous aerobic training & strength training
  Interventions: Behavioral: Vigorous aerobic training
- B: Supervised strength training (Active Comparator): ACTIVE COMPARATOR: Two supervised 45-minute sessions of strength training & Participants will be advised to comply with international recommendations of physical activity (150 min pf MVPA)
  Interventions: Behavioral: Vigorous aerobic training

INTERVENTIONS:
Behavioral: Vigorous aerobic training — Supervised vigorous aerobic training

SUMMARY:
Breast and colon cancer survivors with no evidence of disease, who score less than 45 in the PREDICT questionnaire for fatigue, will be randomized to a supervised strength program versus a supervised resistance program. The primary objective is improvement of cancer-related fatigue.

DETAILED DESCRIPTION:
Patients should have finalized their oncological treatment in the previous 5 years. The sample size (32 patients) was calculated to improve the perception of fatigue score from an anticipated initial 38 to a post-intervention 48.

The control arm consist of supervised strength training in two sessions per week with non-supervised international recommendations for aerobic exercise. The experimental arm will consist of supervised strength + resistance training in two sessions per week.

After evaluating the weekly physical activity through accelerometer, body composition through DEXA and the cardiorespiratory fitness through CPET, participants will initiate the training according to a randomized assignment.

Secondary objectives include:

1. cardiorespiratory fitness,
2. quality of life;
3. adherence to the training program;
4. adherence to international recommendations,
5. body composition,
6. employment status

ELIGIBILITY:
Inclusion Criteria:

* 18-65
* history of breast or colon cancer
* no evidence of disease
* end of treatment in the last five years
* able to understand the questionnaire PERFORM
* able to manage the accelerometer

Exclusion Criteria:

* mobility limitation
* treatment with beta-blockers
* exclusion criteria for CPET

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2016-01; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Improvement in cancer related-fatigue | 4 months

SECONDARY OUTCOMES:
Changes in cardiorespiratory fitness | 4 months
  measured through CPET
Changes in quality of life | 4 months
  measured through EORTC QLQ C30
adherence to the program | 4 months
adherence to international recommendations | 4 months
  measured by accelerometer
Changes in body composition | 4 months
  measured by DEXA (Dual Energy X-Ray Absortiometry)
Employment status | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Itziar Pagola, PhD, Study Director — Universidad Europea de Madrid
Locations (1):
- Hospital Universitario Puerta de Hierro-Majadahonda, Majadahonda, Madrid, Spain